CLINICAL TRIAL: NCT00635986
Title: Analgesic Effect and Plasma Concentration of Epidural Versus Intravenous Fentanyl
Acronym: FTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Adriana Machado Issy/ Professor, Universidade Federal de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fentanyl; No grant
Record Dates: First submitted 2008-01-14; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Fentanyl Analgesia
Keywords: Analgesia; Fentanyl; Orthopedic; Mechanism of action; Surgery
MeSH Terms: conditions — Agnosia | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): group 1 (n = 14) patients received 5 mL of a 100 mcg Fentanyl solution in saline without preservative by the epidural route and 2 mL saline intravenously. Group 2 (n = 15) patients received 5 mL saline by the epidural route and 2 mL (100 mcg) Fentanyl intravenously
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — 100 mcg Fentanyl intravenous or epidural route

SUMMARY:
CONTEXT AND OBJECTIVE: Controversies exist regarding the site of action of Fentanyl after epidural injection. The objective of this investigation was to compare the analgesic effect of epidural and intravenous Fentanyl for lower limb orthopedic surgeries.

DESIGN AND SETTING: A randomized and double-blind study was performed in Hospital São Paulo.

METHODS: 29 patients were divided into two groups. During the postoperative period, in the presence of pain, group 1 (n = 14) patients received 5 mL of a 100 mcg Fentanyl solution in saline without preservative by the epidural route and 2 mL saline intravenously. Group 2 (n = 15) patients received 5 mL saline by the epidural route and 2 mL (100 mcg) Fentanyl intravenously. Analgesic supplementation consisted of 40 mg intravenous Tenoxicam and 5 mL epidural 0.25% bupivacaine (if pain relief was not achieved with Tenoxicam). Pain intensity was evaluated by numerical scale and plasma concentrations of Fentanyl were measured simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Both genders ranging in age from 18 to 65 years, American Society of Anesthesiologists (ASA) Physical Status 1 or 2, scheduled for orthopedic bone surgery of the lower limbs

Exclusion Criteria:

* Patients with infection in the puncture area and coagulation disorders, pregnant patients, and patients using opioids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2005-06 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pain relief | 1 year

SECONDARY OUTCOMES:
fentanyl plasma concentration measure in different times | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Issy, PhD, Study Chair — Federal University of São Paulo

REFERENCES:
- [Derived] Privado MS, Issy AM, Lanchote VL, Garcia JB, Sakata RK. Epidural versus intravenous fentanyl for postoperative analgesia following orthopedic surgery: randomized controlled trial. Sao Paulo Med J. 2010 Jan;128(1):5-9. doi: 10.1590/s1516-31802010000100002. PMID 20512273